CLINICAL TRIAL: NCT05442242
Title: Unicompartmental Knee Arthroplasty vs. High Tibial Osteotomy for Medial Knee Osteoarthritis (UNIKORN): a Study Protocol of a Randomized Controlled Trial
Acronym: UNIKORN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Töölö Hospital (Other)
Responsible Party: Principal Investigator, Juuso Siren, Principal Investigator, Töölö Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/1259/2019
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unicompartmental knee osteoarthritis (Active Comparator)
  Interventions: Procedure: Unicompartmental knee arthroplasty
- High tibial osteotomy (Active Comparator)
  Interventions: Procedure: High tibial osteotomy

INTERVENTIONS:
Procedure: Unicompartmental knee arthroplasty — Medial Unicompartmental knee arthroplasty
  Arms: Unicompartmental knee osteoarthritis
Procedure: High tibial osteotomy — Medial open wedge high tibial osteotomy
  Arms: High tibial osteotomy

SUMMARY:
Unicompartmental knee arthroplasty (UKA) and High Tibial Osteotomy are both valid treatment options for isolated medial knee osteoarthritis. Literature to date is lacking high grade evidence of the outcomes between these procedures. This is a study protocol for randomized controlled trial comparing UKA vs HTO in late stage medial knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Isolated KL 3-4 medial knee arthrosis
* Varus > 3 degrees
* Age 45-65 years

Exclusion Criteria:

* Post-traumatic arthrosis
* Arthrosis in the lateral compartment more than KL grade I in MRI
* Post- traumatic arthrosis
* Instability
* Malignancy Obesity

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
KOOS | 1- year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siren J, Ramo L, Rantasalo M, Komulainen O, Skants N, Reito A, Kosola J, Lindahl J. Unicompartmental knee arthroplasty vs. high tibial osteotomy for medial knee osteoarthritis (UNIKORN): a study protocol of a randomized controlled trial. Trials. 2023 Apr 5;24(1):256. doi: 10.1186/s13063-023-07263-7. PMID 37016454